CLINICAL TRIAL: NCT01393951
Title: Study for Immunogenicity and Safety of ASP7374 for Subcutaneous and Intramuscular Vaccination in Healthy Adults
Brief Title: A Study to Evaluate the Immune Response to the ASP7374 and Its Safety in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7374-CL-0101
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Healthy; Immunogenicity of ASP7374
Keywords: Recombinant Influenza hemagglutinin vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sc dose 1 (Experimental): subcutaneous (sc) vaccination of ASP7374 dose-1
  Interventions: Biological: ASP7374
- sc dose 2 (Experimental): subcutaneous vaccination of ASP7374 dose-2
  Interventions: Biological: ASP7374
- im dose 3 (Experimental): intramuscular (im) vaccination of ASP7374 dose-3
  Interventions: Biological: ASP7374

INTERVENTIONS:
Biological: ASP7374 — subcutaneous and intramuscular

SUMMARY:
This trial is designed as a blinded, randomized and parallel group study to investigate the clinically recommended dosage for ASP7374 based on the comparison of the immunogenicity and safety among two doses of subcutaneous ASP7374 and one dose of intramuscular ASP7374 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: Female: ≥40.0 kg, <70.0 kg, Male: ≥50.0 kg, <80.0 kg
* BMI: ≥17.6, <26.4
* Healthy, as judged by the investigator or sub-investigator based on the results of physical examinations (subjective symptoms and objective findings) and all tests obtained

Exclusion Criteria:

* Scheduled to receive another vaccine during study participation period
* Received influenza vaccine within 180 days prior to the study
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination of the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination of the study vaccine
* Diagnosis of immune deficit in the past, has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome
* Past history of anaphylactic shock or an allergic reaction such as generalized eruption due to food or drug (including vaccines) allergies, fever ≥ 39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* Female subjects who are breastfeeding, pregnant, possibly pregnant, and planning to become pregnant during the study period

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: HI antibody titer | Day 29
Safety: Incidence of Adverse events, vital signs and laboratory tests | 28 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan